CLINICAL TRIAL: NCT06917833
Title: Impact of Maternal Body Mass Index on Infant Hypoxic Events at Time of Delivery ,Cross-sectional Study.
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: MD344/2024
Record Dates: First submitted 2025-03-06; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-02

CONDITIONS: Maternal Obesity; Hypoxia Neonatal
Keywords: maternal obesity; hypoxia neonatal
MeSH Terms: conditions — Pregnancy in Obesity; Asphyxia Neonatorum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- group A (case group ): women with body mass index equal to 25 kg/m2 or more at time of delivery.
  Interventions: Other: compare infant hypoxic events in both groups
- group B ( control group ): women with body mass index (18.5-24.9 kg/m2) at time of delivery
  Interventions: Other: compare infant hypoxic events in both groups

INTERVENTIONS:
Other: compare infant hypoxic events in both groups — early neonatal resuscitation will be done by the pediatrician according to the guidelines, APGAR score of the baby will be calculated,, any hypoxic events will be traced and any need of respiratory support for the baby or NICU admission, as well as weight of the baby, mode of delivery and any birth traumas will be recorded.all this will be compared between two groups.

SUMMARY:
Offspring from overweight or obese mothers appear to be at up to 38% increased risk of being admitted to the neonatal intensive care unit than the offspring of mothers with a normal BMI. In terms of Apgar scores at birth, babies of obese mothers have been reported to have a 31% excess risk of having a low Apgar score (defined at <7 at 1 minute) . Infants born to obese mothers demonstrate a spectrum of outcomes, suggesting that there is a complex interplay of factors that defines the precise altered metabolic environment to which the fetus is exposed and that determines the risk of complications

DETAILED DESCRIPTION:
The investigators need to improve understanding of the specific molecular factors that contribute either individually or synergistically to detrimental fetal outcomes. Moreover, The investigators need to identify the essential maternal markers that need to be tightly regulated during pregnancy to improve outcomes. Here in, The investigators discuss the influence of maternal obesity and factors associated with the obesogenic intrauterine environment on fetal lung development and respiratory outcomes in offspring at birth importantly, The investigators identify a series of molecular changes encountered during pregnancy that may program the observed respiratory outcomes in clinical practice. The effects of maternal obesity on severe neonatal asphyxia may be partly explained by traumatic labor, which often results from macrosomia. Another consequence of maternal obesity is fetal hyperinsulinemia, which may be related to chronic hypoxia even without diabetes . Other mechanisms that explain the effect of maternal obesity on neonatal asphyxia include lipotoxicity, placental inflammation and vasculopathy, and cord coiling. Evidence has demonstrated altered gene expression in full-term newborns of mothers with obesity, involving dysregulation of brain development, inflammatory and immune signaling, glucose and lipid homeostasis, and oxidative stress

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 - 40 years.
2. Term pregnancy (37 weeks gestation or more)
3. Singleton pregnancy
4. Cephalic presentation at time of delivery
5. In labour

Exclusion Criteria:

1. Any medical disorders that affect neonatal outcomes (diabetes mellitus, hypertension, mixed connective tissue disorders)
2. Scarred uterus (myomectomy, previous cesarean section)
3. Macrosomic baby>4 kgs
4. Condition jeopardizing the maternal or fetal life (for example: antepartum hemorrhage, pathological CTG, cord prolapse)
5. Liquor abnormalities (oligohydramnios or polyhydramnios).
6. Other indications for cesarean sections for example: placenta accreta spectrum
7. Smokers.
8. Any abnormalities in follow up of delivery regarding partogram.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant females
Study Population: 18 - 40 years pregnant females 37 weeks or more
Sampling Method: Probability Sample
Enrollment: 544 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2026-01-28 (Estimated); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
Rate of admission to neonatal observation room | 6 hours post delivery

SECONDARY OUTCOMES:
Rate of cesarean-sections. | 12 hours
Oxygen saturation at birth. | 2 hours post delivery
Number of babies with NICU Admission. | 6 hours post delivery
Number of babies with birth trauma. | 2 hours post delivery
Number of babies with meconium aspiration. | 2 hours post delivery